CLINICAL TRIAL: NCT03710655
Title: Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Evaluate the Safety and Efficacy of Apitox Add-on Therapy for Improving Disability and QOL in MS Patients
Brief Title: Evaluate Safety and Efficacy of Apitox Add-on Therapy for Improving Disability and Quality of Life in MS Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Apimeds, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MSKIM10418
Record Dates: First submitted 2018-10-06; First posted 2018-10-18 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Multiple Sclerosis
Keywords: QOL and pain
MeSH Terms: conditions — Multiple Sclerosis; Pain | interventions — Bee Venoms; Histamine

STUDY DESIGN:
Intervention Model Description: 1-1 in two studies of 468 patients total patients 936
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: randomization and blinded personnel at site
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- treatment group (Experimental): skin test, dose escalation, final dose of 1.5mg weekly over 16 weeks of Apitox pure honeybee toxin
  Interventions: Drug: Apitox - pure honeybee toxin
- placebo group (Placebo Comparator): histamine placebo administered intradermally in dose escalation, final dose of 1.5mg weekly over 16 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Apitox - pure honeybee toxin — Intradermal injection of 0.01 microliters
  Other Names: Apitoxin
  Arms: treatment group
Drug: Placebo — Intradermal injection of 0.01 microliters
  Other Names: histamine
  Arms: placebo group

SUMMARY:
Determine the effects of Apitox add-on therapy on the progression of disability in all forms of multiple sclerosis (MS) utilizing the Expanded Disability Status Scale (EDSS) and the MS Functional Composite (MSFC) measure. b. Evaluate the safety and tolerability of add-on Apitox therapy for the treatment of patients with all forms of MS: relapsing-remitting MS (RRMS), primary progressive MS (PPMS) and secondary progressive MS (SPMS). The

DETAILED DESCRIPTION:
The primary efficacy endpoints will assess the effects of Apitox add-on therapy on the changes in EDSS and the MSFC measure from baseline (average Week -1 and Week 1 pre-dose) to Week 16 (Visit 21) versus placebo (histamine). The primary safety endpoint will evaluate, at specified visits, the effects of Apitox add-on therapy on adverse events and tolerability, vital signs, clinical laboratory values, urine pregnancy test, physical exam and 12-Lead ECG. Secondary endpoints will determine the effects of Apitox add-on therapy versus placebo on the improvement in: 1. Quality of life as measured by the MSQoL-54 questionnaire at baseline (average Week -1 and Week 1 pre-dose) and Weeks 3 (Visit 8), Week 10 (Visit 15), Week 15 (Visit 20), Week 16 (Visit 21), Week 17 (Visit 22) and Week 19 (Visit 23). 2. Ambulatory and functional disability as measured by the individual Functional System Scores (FSS) at baseline (average Week -1 and Week 1 pre-dose) and Visits 8, 15, 20, 21, 22 and 23. 3. Progression of disability utilizing the change in EDSS and MSFC obtained at baseline (average Week -1 and Week 1 1 pre-dose) and Visits 8, 15, 20, 21, 22 and 23. 3. Progression of disability utilizing the change in EDSS and MSFC obtained at baseline (average Week -1 and Week 1 pre-dose) and assessed at and Visits 8, 15, 20, 22 and 23. 4. Pain and physical function as assessed with the Pain Intensity Numerical Rating Scale (PI-NRS) and Patient Global Impression of Change (PGIC) at baseline (average Week -1 and Week 1 pre-dose) and Visits 8, 15, 20, 21, 22 and 23. 5. Disease status using Patient Global Assessment (PGA), and Physician's Global Assessment (PhGA) at baseline (average Week -1 and Week 1 pre-dose) and Visits 8, 15, 20, 21, 22 and 23. Exploratory endpoints will assess, in a subset of subjects, changes in MS lesions from baseline (Week -2 or within the past 52 weeks) . Prior to randomization, subjects will undergo a skin test with Apitox (50 micrograms) to exclude those with systemic hypersensitivity to the product. Subjects will continue taking their regular MS treatments throughout the study. During the study, subjects will receive an additional 1 gram ascorbic acid per day and must not consume alcohol. After a screening period of up to 3 weeks, approximately 436 eligible subjects will be randomized in a 1:1 ratio to either Apitox (n=218) or Placebo (n=218). The fixed histamine placebo dosage was designed to be sub-therapeutic and mimic the sensation of a bee sting. All injections will be administered intradermally according to the schedule and anatomical sites provided in Appendix 1, twice weekly for 3 weeks, and then once weekly for another 12 weeks. Each subject's starting dose will be 0.2 mL (Week 1; Visit 3) and will be escalated at every visit in 0.2 mL increments up to the maximum dose of 1.5 mL (1500 micrograms at Week 4; Visit 9). At Visits 9 through 20, subjects will continue to receive 1.5 mL Apitox or placebo for the rest of the study. A subset of the randomized subjects (n=44) will undergo MRI testing for exploratory analyses of changes in MS lesions at follow-up Visit 21 (Week 16). There are 3 follow up visits (Visits 21, 22 and 23) at 1, 2 and 4 weeks post-treatment after the last maximum dose visit (Week 15; Visit 20). During treatment, visits should be at least 3 days apart. The duration of the study is up to 22 weeks that includes up to 3 weeks of screening, 15 weeks on treatment, and 4 weeks for follow-up visits. If a subject experiences an exacerbation of MS during the study, he or she should inform the site as soon as possible. The subject's primary care physician will be consulted if appropriate additional treatment can be performed at the site; e.g. intravenous (IV) corticosteroids. The primary care physician and PI will determine if the subject will continue in the trial. If the subject is discontinued, she or he will have an early termination (ET) visit. If a subject experiences an immediate or delayed hypersensitivity reaction from Apitox or histamine study treatments, the subject will undergo emergency procedures described in Sections 5.4.5 and 5.4.6. Dosing will be carried out at clinical sites in geographical areas with access to emergency facilities (i.e., near hospital or clinic with an Emergency Care Facility). Each site has personnel trained in emergency response including cardiopulmonary resuscitation (CPR), and each has rescue parenteral epinephrine available. Before discharge at Week 1 (Visit 3), each subject will be provided epinephrine for the treatment of anaphylactic shock (e.g. EpiPen® Auto-Injector) and will be advised that this should always be available to them. In the event of a severe anaphylactic reaction, subjects will stop Apitox therapy and will be discontinued from the study. This study will be monitored by a Safety Monitoring Committee (SMC). The SMC will be comprised of an independent physician, the Medical Monitor and the Investigator. The independent physician is not directly affiliated with the protocol under review. The SMC will meet to review the safety of subjects who participate in the trial and will meet, if required, to advise the sponsor if enrollment and dose escalation should continue for a specific subject

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have provided written informed consent and authorization for disclosure of protected health information must meet the following criteria:

  1. Men or women aged 18 to 65 years inclusive.
  2. Confirmed diagnosis of MS as defined by the McDonald criteria [25].
  3. Receiving disease modifying treatment and/or treatment for symptoms of MS at baseline. Subjects will be allowed to continue their MS treatment regimens throughout the trial (see Sections 7.4 and 7.5 for prior and allowed medications, respectively, during the trial).
  4. Females of childbearing potential must be willing to use an acceptable method of contraception. A woman is considered of childbearing potential if she is not surgically sterile or if her last menstrual period was <12 months prior to Visit 1. Acceptable methods of contraception for this study include surgical sterilization, oral or depot contraceptives (taken for at least 60 days before Week 1), intrauterine devices, diaphragm with spermicide, or other methods on a subject-by-subject basis.
  5. Baseline EDSS score of 0.0-6.0 (average Week -1 and Week 1 pre-dose).
  6. Able to understand and be willing to comply with all study requirements, particularly the regimen for administration of investigational product.

Exclusion Criteria:

* Any subject who meets any of the following criteria will not qualify for entry into the study:

  1. A history of allergic reactions or drug hypersensitivity to honeybee venom.
  2. A systemic reaction to a skin test for hypersensitivity to Apitox. Phase 3 Trial Evaluating the Safety and Efficacy of Apitox Add-on Therapy Protocol 02-2014 for Improving Disability and Quality of Life in Patients with Multiple Sclerosis 07 April 2017
  3. History of abnormal MRI scan, not attributable to MS.
  4. Neurological disorder other than MS, acute or chronic infection.
  5. Malignant neoplasm or metastasis except for basal and squamous skin cancers.
  6. Coronary artery disease or prior myocardial infarction.
  7. Use of beta-blockers, drugs considered potent CYP450 inhibitors (see a list of moderate and strong CYP450 inhibitors in Appendix 9), alcohol, or preparations containing histamine (such as Prokarin™) during the study period.
  8. Insulin dependent diabetes mellitus or unstable type 2 diabetes mellitus.
  9. Any clinically significant ECG abnormalities (e.g. ischemic changes), as determined by the Investigator.
  10. Any abnormal clinical or laboratory parameter that is considered clinically significant or has Grade 3 or higher as specified in the "Guidance for Industry - Toxicity Grading Scales for Healthy Adult and Adolescent Volunteers enrolled in Preventative Vaccine Clinical Trials" (Appendix 8). Subjects with abnormal hepatic and renal labs that are considered mild (Grade 1) or moderate (Grade 2) and not clinically significant (Appendix 8) will be monitored during the trial. 11. Recent (within 1 year of screening) alcohol abuse or use of marijuana or illicit drugs.

  12. Females who are lactating/breastfeeding or who plan to breastfeed while on study through 2 weeks after receiving the last dose of study drug.

  13. Females who are pregnant or who plan to become pregnant. 14. Use of an investigational product within a period of 28 days prior to enrollment in the study that would, in the opinion of the Investigator, confound the treatment for QoL or pain reduction.

  15. Any condition that, in the opinion of the Investigator, would place the subject at increased risk or may confound the study results. DOSAGE

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 468 (Estimated)
Dates: Start 2019-04 (Estimated); Primary Completion 2019-08 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Expanded Disability Status Scale (EDSS) | 16 weeks
MS Functional Composite (MSFC) | 16 weeks

SECONDARY OUTCOMES:
Quality of life questionnaire (MSQoL-54) | 16 weeks
Functional System Scores (FSS) | 16 weeks
Pain Intensity Numerical Rating Scale (PI-NRS) | 16 weeks
Patient Global Impression of Change (PGIC) | 16 weeks
Patient Global Assessment (PGA) | 16 weeks
Physician's Global Assessment (PhGA) | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Robert Brooks, PhD, Study Director — Apimeds, Inc.

IPD SHARING:
Plan to Share IPD: Undecided